CLINICAL TRIAL: NCT04847050
Title: A Trial of the Safety and Immunogenicity of the COVID-19 Vaccine (mRNA-1273) in Participants With Hematologic Malignancies and Various Regimens of Immunosuppression, and in Participants With Solid Tumors on PD1/PDL1 Inhibitor Therapy, Including Booster Doses of Vaccine
Brief Title: A Trial of the Safety and Immunogenicity of the COVID-19 Vaccine (mRNA-1273) in Participants With Hematologic Malignancies and Various Regimens of Immunosuppression, and in Participants With Solid Tumors on PD1/PDL1 Inhibitor Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Gulley, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10000115; 000115-C
Record Dates: First submitted 2021-04-14; First posted 2021-04-15 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor Malignancy; Hematologic Malignancy; Leukemia; Lymphoma; Multiple Myeloma
Keywords: mRNA-1273 vaccine; moderna; SARS-CoV-2; booster shot
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Multiple Myeloma | interventions — RNA, Messenger; 2019-nCoV Vaccine mRNA-1273; Electrocardiography; Anti-Bacterial Agents; Antifungal Agents; Antiemetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 messenger ribonucleic acid (mRNA) (Experimental): 100 mcg (0.5 mL) messenger ribonucleic acid (mRNA)-1273 injection intramuscular (IM) on days 1 and 29; with option for subsequent booster dose(s), 100 mcg (0.5 mL) mRNA-1273 injection (IM) no less than 4 weeks after day 29
  Interventions: Biological: Messenger ribonucleic acid (mRNA)-1273 Vaccine; Biological: Messenger ribonucleic acid (mRNA)-1273 Vaccine Booster; Diagnostic Test: ECG; Other: Antibiotics; Other: Anti-viral agents; Other: Anti-fungal agent; Other: Anti-emetics
- Arm 2 messenger ribonucleic acid (mRNA) (Experimental): 100 micrograms (0.5 mL) messenger ribonucleic acid (mRNA) injection on day (D)1
  Interventions: Biological: Messenger ribonucleic acid (mRNA)-1273 Vaccine; Diagnostic Test: ECG; Other: Antibiotics; Other: Anti-viral agents; Other: Anti-fungal agent; Other: Anti-emetics

INTERVENTIONS:
Biological: Messenger ribonucleic acid (mRNA)-1273 Vaccine — A rapid response, proprietary messenger RNA (mRNA)-based vaccine platform. 100 mcg administered intramuscular (IM) on Day 1 and 29 for vaccine naive cohorts.
  Other Names: mRNA-1273
Biological: Messenger ribonucleic acid (mRNA)-1273 Vaccine Booster — A rapid response, proprietary messenger RNA (mRNA)-based vaccine platform. 100 mcg administered intramuscular (IM) on Day 1 for vaccine booster cohorts. Participants may receive up to 3 booster injections on study.
  Other Names: mRNA-1273
  Arms: Arm 1 messenger ribonucleic acid (mRNA)
Diagnostic Test: ECG — Baseline (-28 days/Day 1); and Day 29 (+/- 3 days).
  Other Names: Electrocardiogram
Other: Antibiotics — Use of prophylactic antibiotics is recommended according to institutional standards.
Other: Anti-viral agents — Use of prophylactic antiviral agents is recommended according to institutional standards.
Other: Anti-fungal agent — Use of prophylactic antifungal agents is recommended according to institutional standards.
Other: Anti-emetics — Use of prophylactic anti-emetics is recommended according to institutional standards.

SUMMARY:
Background:

Coronavirus disease (COVID-19) is a viral infection. It has spread rapidly across the globe. It has overwhelmed health systems. Researchers are concerned that it may undo years of progress in the reduction of cancer-specific death. They want to test a vaccine that might protect people with cancer from COVID-19.

Objective:

To test the safety and efficacy of a vaccine using messenger ribonucleic acid (mRNA)-1273 that may protect people with cancer from COVID-19.

Eligibility:

Adults ages 18 and older who have a solid tumor or blood cancer and who may benefit from a vaccine that might prepare their immune system for fighting and preventing infection from COVID-19. Patients with solid tumors must be receiving treatment with an immunotherapy agent.

Design:

Participants will be screened with a medical history, medicine review, and physical exam. They will have blood tests. They will have a pregnancy test if needed.

Participants will get 2 doses of the mRNA-1273 vaccine if they have not been vaccinated already. It will be injected into a muscle in the arm on Days 1 and 29. They will be followed for 12 months after the second dose.

Participants will have study visits at the Clinical Center on Days 1, 29, 36,57, 209, and 394. Some visits will last about 4-6 hours. Patients will be able to get up to 3 doses of mRNA-1273 as a booster on trial if they have already completed a primary series of a vaccine. Participants who have already received a booster dose of vaccine will be able to enroll to receive additional boosters. It will be injected into a muscle in the arm on Day 1. Participants will be followed for 12 months after their last booster injection. Participants who receive booster doses will have study visits at the Clinical Center on Days 1, 29, 57, 180 and 360.

Participants will give blood and saliva samples for research.

Participation will last about 16 months.

DETAILED DESCRIPTION:
Design of the Study:

This is an open-label, multicenter clinical trial designed to evaluate the safety, reactogenicity and primary immunogenicity of the messenger ribonucleic acid (mRNA)-1273 vaccine administered in 2 doses, 28 days apart, in participants who have hematological malignancy and are immunosuppressed due to their disease and/or treatment or receiving a Programmed cell death protein 1 (PD-1)/Programmed death-ligand 1 (PDL-1) inhibitor for treatment of a solid tumor can be associated with appropriately high rates of development of neutralizing antibodies of mRNA-1273. The trial will also evaluate the safety, reactogenicity and immunogenicity after administration of additional booster doses of the vaccine.

Study Phase:

Study Population:

For the vaccine-na(SqrRoot) ve cohorts, up to 80 participants will be enrolled.

* 20 participants with solid tumor malignancies who have initiated PD1/PDL1 inhibitor therapy as part of standard of care and are deemed to have a stable regimen without the need for any immunosuppressive therapy or corticosteroids.
* 60 participants with leukemia, lymphoma, multiple myeloma and participants post-allogeneic stem cell transplant will be enrolled based on their perceived risk of immunosuppression.

For the previously-vaccinated (also known as "booster") cohorts, up to 140 participants will be enrolled for booster injections. All participants on the vaccine-na(SqrRoot) ve cohorts will have the option of receiving boosters; however, they will not count towards the maximum accrual goal for each of the booster groups. Note: All participants will be eligible to receive up to three (3) booster doses of vaccine on study.

* 20 participants with solid tumor malignancies who have initiated PD1/PDL1 inhibitor therapy as part of standard of care and are deemed to have a stable regimen without the need for any immunosuppressive therapy or corticosteroids.
* 20 participants with chronic lymphocytic leukemia who are not currently on any therapies
* 20 participants with chronic lymphocytic leukemia who are on Bruton's tyrosine kinase (BTK) inhibitor therapy alone
* 30 participants with any chimeric antigen receptor (CAR) T Cell therapy for a hematologic malignancy
* 20 participants post-allogeneic stem cell transplant
* 20 participants with other hematologic malignancies
* Up to 10 participants with any solid tumor who are not otherwise eligible for any of the other cohorts

Number of Sites: 2

Description of Study Product or Intervention:

mRNA-1273 Injection (Drug Product) is an lipid nanoparticles (LNPs) dispersion containing a single mRNA sequence (Drug Substance) that encodes the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) S glycoprotein stabilized in the prefusion conformation. The mRNA-1273 Drug Substance is combined with a mixture of 4 lipids common to the Moderna's mRNA vaccine platform: SM-102 (a custom-manufactured, ionizable lipid) and 3 commercially available lipids, cholesterol, distearoylphosphatidylcholine (DSPC), and 1,2-dimyristoyl-rac-glycero-3-methoxypolyethylene glycol-2000 (PEG2000-DMG) (https://doi.org/10.1038/s41587-020- 00807-1). mRNA-1273 Injection is provided as a sterile solution for injection, white to off white dispersion in appearance.

Presentation: mRNA-1273 Injection is provided as a sterile solution for injection at a concentration of 0.2 mg/mL in 20 mM trometamol (Tris) buffer containing 87 mg/mL sucrose and 4.3 mM acetate, at potential hydrogen (pH) 7.5. mRNA-1273 Injection is presented in 10R USP Type I borosilicate glass vials with PLASCAP vial seal containing a 20 mm FluroTec-coated plug stopper and has a 6.3 mL nominal fill volume. This vial may be used for more than one participant.

mRNA-1273 Injection must be stored frozen at -15 degrees C to -25 degrees C until thawed for use and then stored refrigerated at 2 degrees C to 8 degrees C for up to 30 days (once thawed it must not be refrozen)

Each dose of 100 mcg (0.5 mL) will be administered via IM injection into the deltoid muscle on Days 1 and 29 (+/- 3 days) for the vaccine-na(SqrRoot) ve cohorts. Up to 3 additional (booster) doses of the vaccine may also be administered.

Study Objectives:

Primary:

* To evaluate the safety and reactogenicity of the mRNA-1273 vaccine administered in 2 doses, 28 days apart, in participants who have a hematological malignancy and are immunosuppressed due to their disease and/or treatment, or receiving a PD-1/PDL-1 inhibitor for treatment of a solid tumor for patients who are vaccine-na(SqrRoot) ve
* To evaluate the safety and reactogenicity of booster doses of mRNA-1273 vaccine administered to participants who have previously received an mRNA or alternative vaccine regimen
* To evaluate the safety and reactogenicity of booster doses of mRNA-1273 administered to participants with chronic lymphocytic leukemia (CLL) who are either off treatment or are engaging in a 3-week BTK inhibitor interruption to enhance vaccine immunogenicity
* To assess the immunogenicity of mRNA-1273 in participants with cancer, as assessed by the titer or level of specific binding antibody (bAb)

Secondary:

* To evaluate the immunogenicity of the mRNA-1273 vaccine administered in 2 doses 28 days apart, as assessed by the titer or level of neutralizing antibody (nAb) in the vaccine-na(SqrRoot) ve cohorts
* To evaluate the immunogenicity of booster doses of mRNA-1273 vaccine administered to participants who have previously been vaccinated against SARS-CoV2 with any prior vaccine regimen. as assessed by the titer or level of neutralizing antibody (nAb)

Exploratory:

* To assess immune responses against the SARS-CoV-2 nucleocapsid and spike proteins
* To evaluate salivary measurement of immunoglobulin G (IgG) antibodies against the SARS-CoV-2 nucleocapsid and spike (S) proteins

Duration of Individual Participant Participation:

The duration for each individual participation is approximately 14 months (from first contact to last visit).

Study Duration:

Study duration is anticipated to be 16 months (from start of screening to last Participant/last visit).

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must meet all the inclusion criteria in order to be eligible to participate in the study.

Participants must have one of the following:

* Histologically or cytologically confirmed solid tumor receiving a standard of care programmed cell death protein 1 (PD1)/Programmed death-ligand 1 (PDL1) inhibitor for treatment of their solid tumor (inclusive of Hodgkin Lymphoma and Primary Mediastinal B-Cell Lymphoma participants receiving PD1/PDL1 inhibitors as standard of care therapy)
* Confirmed diagnosis of acute leukemia (myeloid (AML) or lymphoid (ALL) or other acute leukemia; multiple myeloma; Waldenstrom macroglobulinemia
* Confirmed diagnosis of lymphoma, including small lymphoblastic lymphoma (i.e.,chronic lymphocytic leukemia)

  * Be post allogeneic stem cell transplantation (for any indication)
  * Be an adult patient (aged 18 or older) with any malignancy who does not fit any of the above categories
  * Age >=18 years.
  * History of adequate organ and marrow function on a recent laboratory assessment (within 4 weeks of administration of vaccine), as defined below:
* Absolute lymphocyte count-Minimum value of 200 cells per mcL
* Absolute neutrophil count-Minimum value of 500 cells per mcL
* Platelets-Minimum value of 25,000 cells per mcL
* Total bilirubin-Maximum value of 3.0 x upper limit of normal
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine transaminase ALT serum glutamic-pyruvic transaminase (SGPT)-Maximum value of 5.0 x upper limit of normal
* Creatinine-Maximum value of 3.0 x upper limit of normal (if elevated, use of creatinine calculated clearance will be necessary, as below)
* Creatinine clearance (only necessary for participants with elevated creatinine)-For participants with Chronic Kidney Disease, a calculated

Glomerular Filtration Rate minimum will be required as follows: >30 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal.

* Participants with history of human immunodeficiency virus (HIV) may enroll
* Participants with history of chronic hepatitis B virus (HBV) must be on suppressive therapy (if indicated) with undetectable viral load.
* Participants with a known history of hepatitis C virus (HCV) infection must have been treated and cured with an undetectable HCV viral load. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* A negative urine/serum pregnancy test for females of childbearing potential. The effects of mRNA-1273 Vaccine on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for 30 days after the last study treatment.

Note: A female is considered to be of childbearing potential if she has experienced menarche and is not permanently sterile (i.e., hysterectomy, bilateral oophorectomy, or tubal ligation) or postmenopausal (postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause and with a serum follicle-stimulating hormone test result in the postmenopausal range).

Effective methods of contraception:

* Intrauterine device.
* Stable dose of hormonal birth control, such as those listed below, for at least 3 months prior to enrollment.

  * Hormonal contraceptive tablets.
  * Injectable hormonal contraceptives.
  * Implanted hormonal contraceptives.
  * Cutaneous contraceptive patches.
  * Intravaginal hormonal contraceptive rings.

At least 1 barrier method. Effective barrier methods for use in this study are:

* Male or female condom.
* Diaphragm.
* Creams or gels that contain a chemical to kill sperm

If a female patient has a male participant who has had surgery to prevent pregnancy (vasectomy), that will be considered evidence of effective contraception.

* Ability to understand and the willingness to sign a written informed consent document.
* CLL participants undergoing Bruton tyrosine kinases inhibitors (BTKi) treatment interruption: Must be receiving treatment with a BTKi for 6 months prior to vaccination and be willing to hold their treatment for up to 3 weeks around the time of vaccination.

EXCLUSION CRITERIA:

All participants meeting any of the exclusion criteria at baseline will be excluded from study participation.

* Within 14 days of known exposure to someone with confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection or coronavirus disease (COVID-19).
* Acutely ill or febrile 24 hours prior to or at the Screening Visit (Day 0). Fever is defined as a body temperature greater than or equal to 38.0 degrees C/100.4 degrees F. Participants meeting this criterion may be rescheduled within the relevant window periods. Afebrile participants with minor illnesses can be enrolled at the discretion of the investigator.
* Participants on the vaccine na(SqrRoot) ve arms cannot have received any doses of the COVID-19

vaccine.

Participants who have not completed a standard vaccination series due to initiation of vaccination in a foreign location (e.g., single dose of Astra-Zeneca vaccine or a similar situation) may be enrolled after discussion with the principal investigator.

Participants on the booster arms must have received all doses of their initial COVID-19 vaccine (Participants vaccinated with the Janssen vaccine must have received the single dose of that Emergency Use Authorization (EUA) vaccine for COVID19, but all others must have received 2 doses) at least 4 weeks prior to vaccination on protocol. Participants will be allowed to enroll if they have already received booster doses of vaccine prior to enrolling on the protocol at least four weeks prior to vaccination on protocol. In this case, the protocol will administer a single booster dose of vaccination. Documentation will be required.

* Known diagnosis of chronic pulmonary disease (e.g., chronic obstructive pulmonary disease, asthma) that is not controlled.
* Chronic cardiovascular disease that is not controlled.
* Participants with a history of myocarditis (inflammation of the heart) or pericarditis (inflammation of the pericardium)
* History of anaphylaxis, urticaria, or other significant adverse reaction requiring medical intervention after receipt of a vaccine.
* Bleeding disorder considered a contraindication to intramuscular (IM) injection or phlebotomy.
* Participated in an interventional clinical trial with an investigational agent within 28 days prior to the Screening Visit (Day 0) or plans to do so while participating in this study. The site investigator may enroll a participant on the trial earlier than 28 days if enough time has passed to ensure that at least five half-lives have occurred.
* Prior/Concomitant Therapy

  * Has received prior radiotherapy within 14 days before the first dose of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 7-day washout is permitted for palliative radiation (less than or equal to 2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
  * Has received a live vaccine within 30 days before the first dose of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist (registered trademark)) are live attenuated vaccines and are not allowed.
  * Has received an inactivated vaccine within 14 days before the first dose of study treatment.
* Have major surgical procedures within 28 days or non-study-related minor procedures within 7 days before the first dose of study treatment. In all cases, the participant must be sufficiently recovered and stable before treatment administration.

  --History of severe allergic reactions to any components of the study treatment.
* Has uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, severe or ongoing interstitial lung disease (ILD), serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs), or compromise the ability of the participant to give written informed consent.
* Active tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice).
* History of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has involvement in the planning and/or conduct of the study.
* Female who is pregnant or breastfeeding
* Male or female participant of reproductive potential who are not willing to employ effective birth control from screening to 30 days after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000115-C.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in the following groups: Chronic Lymphocytic Leukemia (CLL) Not on Active Therapy - Booster Phase; Chronic Lymphocytic Leukemia(CLL) Receiving Bruton´s Tyrosine Kinase(BTK) Interruption-Booster Phase; Chimeric Antigen Receptor (CAR) T Cell Therapy - Booster Phase; and Other Adult Solid Tumor - Booster Phase. In the initial phase, 15 participants started & 4 started in the booster phase = 19 participants enrolled. Participants who crossed over are noted in the table.
Groups:
- Hematologic Low Immunosuppression - Initial Phase; Hematologic Intermediate Immunosuppression - Initial Phase; Hematologic High Immunosuppression - Initial Phase; Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Initial Phase: 100 mcg (0.5 mL) messenger ribonucleic acid (mRNA)-1273 injection, intramuscular (IM) on days 1 and 29; with option for subsequent booster dose, 100 mcg (0.5 mL) mRNA-1273 injection (IM) no less than 4 weeks after day 29.
- Chronic Lymphocytic Leukemia (CLL) Not on Active Therapy - Booster Phase; Chronic Lymphocytic Leukemia(CLL) Receiving Bruton´s Tyrosine Kinase(BTK) Interruption-Booster Phase; Chimeric Antigen Receptor (CAR) T Cell Therapy - Booster Phase; Other Adult Solid Tumor - Booster Phase: No participants were enrolled in this group.
  100 mcg (0.5 mL) messenger ribonucleic acid (mRNA)-1273 injection on day (D)1.
- Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Booster Phase; Post Allogeneic Transplant - Booster Phase: 100 mcg (0.5 mL) messenger ribonucleic acid (mRNA)-1273 injection on day (D)1.
- Other Hematologic Malignancy - Booster Phase: 100 mcg (0.5 mL) messenger ribonucleic acid (mRNA)-1273 injection, intramuscular (IM) on day 1.
Period: Initial Phase
Arm/Group | Hematologic Low Immunosuppression - Initial Phase | Hematologic Intermediate Immunosuppression - Initial Phase | Hematologic High Immunosuppression - Initial Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Initial Phase | Chronic Lymphocytic Leukemia (CLL) Not on Active Therapy - Booster Phase | Chronic Lymphocytic Leukemia(CLL) Receiving Bruton´s Tyrosine Kinase(BTK) Interruption-Booster Phase | Chimeric Antigen Receptor (CAR) T Cell Therapy - Booster Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Booster Phase | Post Allogeneic Transplant - Booster Phase | Other Hematologic Malignancy - Booster Phase | Other Adult Solid Tumor - Booster Phase
Started | 2 | 3 | 7 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participants Eligible for the Booster Phase (All participants will be eligible to receive up to (3) booster doses of vaccine on study.) | 1 | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 3 | 7 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Booster Phase
Arm/Group | Hematologic Low Immunosuppression - Initial Phase | Hematologic Intermediate Immunosuppression - Initial Phase | Hematologic High Immunosuppression - Initial Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Initial Phase | Chronic Lymphocytic Leukemia (CLL) Not on Active Therapy - Booster Phase | Chronic Lymphocytic Leukemia(CLL) Receiving Bruton´s Tyrosine Kinase(BTK) Interruption-Booster Phase | Chimeric Antigen Receptor (CAR) T Cell Therapy - Booster Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Booster Phase | Post Allogeneic Transplant - Booster Phase | Other Hematologic Malignancy - Booster Phase | Other Adult Solid Tumor - Booster Phase
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 10 | 0
Number of Participants Who Crossed Over From Hematologic Low Immunosuppression -Initial Phase (Ph) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Number of Participants Who Crossed Over From Hematologic Intermediate Immunosuppression Initial Ph. | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Number of Participants Who Crossed Over From Hematologic High Immunosuppression -Initial Phase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Number of Participants Who Crossed Over From Solid Tumor on PD1/PDL-1 -Initial Phase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 10 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hematologic Low Immunosuppression - Initial Phase | Hematologic Intermediate Immunosuppression - Initial Phase | Hematologic High Immunosuppression - Initial Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Initial Phase | Other Hematologic Malignancy - Booster Phase | Total
Number analyzed (Participants) | 2 | 3 | 7 | 3 | 4 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 6 | 2 | 2 | 13
  >=65 years | 0 | 2 | 1 | 1 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.85 (10.54) | 62.96 (7.7) | 49.51 (16.42) | 59.17 (9.8) | 62.38 (13.81) | 56.01 (13.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 1 | 0 | 5
  Male | 0 | 2 | 6 | 2 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 7 | 2 | 4 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 3 | 2 | 0 | 7
  White | 1 | 2 | 3 | 0 | 4 | 10
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 7 | 3 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grades 1-5 Solicited (Expected) and/or Unsolicited (Unexpected) Adverse Events (AE's): Initial Phase
Description: Solicited (expected) local and systemic Adverse Reactions (ARs) through 7 days after each injection were assessed using the clinical abnormalities section of the Food and Drug Administration (FDA) -Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. Unsolicited (unexpected) adverse events (AEs) through 28 days after each injection and serious adverse events (SAE's) throughout the entire study period were assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: 7 and 28 days after each injection and throughout the entire study period, a median of 19.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hematologic Low Immunosuppression - Initial Phase | Hematologic Intermediate Immunosuppression - Initial Phase | Hematologic High Immunosuppression - Initial Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Initial Phase
Number analyzed (Participants) | 2 | 3 | 7 | 3
Participants
  Grade 3 Serious Unsolicited -Immune system disorders - Other, GVHD | 0 | 0 | 1 | 0
  Grade 3 Serious Unsolicited - Pneumothorax | 0 | 0 | 0 | 1
  Grade 1 Non-serious Solicited - Anal hemorrhage | 0 | 0 | 1 | 0
  Grade 1 Non-serious Solicited - Constipation | 0 | 0 | 1 | 0
  Grade 1 Non-serious Solicited - Cough | 1 | 0 | 1 | 0
  Grade 1 Non-serious Solicited - Hemorrhoidal hemorrhage | 0 | 0 | 1 | 0
  Grade 1 Non-serious Solicited - Hypertension | 0 | 1 | 2 | 2
  Grade 1 Non-serious Solicited - Hypoalbuminemia | 0 | 0 | 1 | 0
  Grade 1 Non-serious Solicited - Hypokalemia | 0 | 0 | 1 | 0
  Grade 1 Non-serious Solicited - Infections and Infestations - Other, GI Virus | 0 | 0 | 1 | 0
  Grade 1 Non-serious Solicited - Nasal congestion | 0 | 0 | 1 | 0
  Grade 1 Non-serious Solicited - White blood cell decreased | 0 | 0 | 1 | 0
  Grade 1 Non-serious Solicited - Arthralgia | 0 | 0 | 1 | 0
  Grade 1 Non-serious Solicited - Dyspnea | 1 | 0 | 0 | 0
  Grade 1 Non-serious Solicited - Weight gain | 0 | 0 | 0 | 0
  Grade 2 Non-serious Solicited - Anorexia | 0 | 0 | 1 | 0
  Grade 2 Non-serious Solicited - Blurred vision | 0 | 0 | 1 | 0
  Grade 2 Non-serious Solicited - Conjunctivitis | 0 | 0 | 2 | 0
  Grade 2 Non-serious Solicited - Creatinine clearance | 0 | 0 | 1 | 0
  Grade 2 Non-serious Solicited - Dry mouth | 0 | 0 | 1 | 0
  Grade 2 Non-serious Solicited - Dysgeusia | 0 | 0 | 1 | 0
  Grade 2 Non-serious Solicited - Hypotension | 0 | 0 | 1 | 0
  Grade 2 Non-serious Solicited - Immune system disorders - Other, GVHD | 0 | 0 | 1 | 0
  Grade 2 Non-serious Solicited - Lymphocyte count decreased | 0 | 0 | 1 | 0
  Grade 2 Non-serious Solicited - Rash maculopapular | 0 | 0 | 1 | 0
  Grade 2 Non-serious Solicited - Upper respiratory infection | 0 | 0 | 1 | 0
  Grade 2 Non-serious Solicited - Viremia | 0 | 0 | 1 | 0
  Grade 2 Non-serious Solicited - Infections and infestations - Other, COVID | 1 | 0 | 1 | 0
  Grade 2 Non-serious Solicited - Neutrophil count decreased | 1 | 0 | 0 | 0
  Grade 2 Non-serious Solicited - Pneumonitis | 1 | 0 | 0 | 0
  Grade 2 Non-serious Solicited - Cough | 0 | 0 | 0 | 1
  Grade 2 Non-serious Solicited - Dental caries | 0 | 0 | 0 | 1
  Grade 2 Non-serious Solicited - Dyspnea | 0 | 0 | 0 | 1
  Grade 2 Non-serious Solicited - Hypothyroidism | 0 | 0 | 0 | 1
  Grade 2 Non-serious Solicited - Non-cardiac chest pain | 0 | 0 | 0 | 1
  Grade 2 Non-serious Solicited - Pneumothorax | 0 | 0 | 0 | 1
  Grade 2 Non-serious Solicited - Weight gain | 0 | 0 | 0 | 1
  Total Non-serious Solicited | 0 | 0 | 0 | 0
  Total Serious Solicited | 0 | 0 | 0 | 0
  Total Non-serious Unsolicited | 2 | 1 | 7 | 2
  Total Serious Unsolicited | 0 | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Reactogenicity of Messenger Ribonucleic Acid (mRNA)-1273 Vaccine: Initial Phase
Description: Reactogenicity of mRNA-1273 vaccine was assessed by physical examination findings following vaccination. A physical exam will be performed to assess general physical condition in the following areas: supraclavicular and axillary lymph nodes, cardiovascular, pulmonary, abdomen and skin and include an assessment of pain, tenderness, erythema, induration and warmth at the injection site, fever, chills, arthralgia/joint pain, malaise/fatigue, myalgia/body aches, headache, nausea, vomiting, and abdominal pain following vaccination.
Time Frame: End of 15-minute observation period following each vaccination on Day 1 and Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Hematologic Low Immunosuppression - Initial Phase | Hematologic Intermediate Immunosuppression - Initial Phase | Hematologic High Immunosuppression - Initial Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Initial Phase
Number analyzed (Participants) | 2 | 3 | 7 | 3
Participants
  Day 1 - Pain | 2 | 2 | 6 | 3
  Day 1 - Tenderness | 1 | 2 | 3 | 0
  Day 1 - Erythema | 1 | 0 | 2 | 0
  Day 1 - Induration and warmth at the injection site | 0 | 0 | 3 | 1
  Day 1 - Fever | 0 | 0 | 0 | 0
  Day 1 - Chills | 0 | 0 | 1 | 0
  Day 1 - Arthralgia/joint pain | 0 | 0 | 0 | 0
  Day 1 - Malaise/fatigue | 1 | 0 | 2 | 0
  Day 1 - Myalgia/body aches | 1 | 0 | 2 | 0
  Day 1 - Headache | 0 | 0 | 2 | 0
  Day 1 - Nausea | 0 | 0 | 0 | 0
  Day 1 - Vomiting | 0 | 0 | 0 | 0
  Day 1 - Abdominal pain | 0 | 0 | 0 | 0
  Day 29 - Pain | 2 | 2 | 5 | 3
  Day 29 - Tenderness | 2 | 1 | 4 | 1
  Day 29 - Erythema | 0 | 0 | 2 | 0
  Day 29 - Induration and warmth at the injection site | 1 | 1 | 3 | 1
  Day 29 - Fever | 0 | 0 | 0 | 0
  Day 29 - Chills | 0 | 0 | 1 | 1
  Day 29 - Arthralgia/joint pain | 1 | 0 | 0 | 0
  Day 29 - Malaise/fatigue | 0 | 0 | 5 | 1
  Day 29 - Myalgia/body aches | 1 | 0 | 3 | 3
  Day 29 Headache | 1 | 1 | 3 | 2
  Day 29 - Nausea | 0 | 0 | 1 | 0
  Day 29 - Vomiting | 0 | 0 | 0 | 0
  Day 29 - Abdominal pain | 0 | 0 | 0 | 0
  Day 1- Hypertension | 0 | 0 | 0 | 0
  Day -29 Systolic Hypertension | 0 | 2 | 4 | 0

3. Primary Outcome: Number of Participants With Grades 1-5 Solicited (Expected) and/or Unsolicited (Unexpected) Adverse Events (AE's): Booster Phase
Description: as for outcome 1
Time Frame: 7 and 28 days after each injection and throughout the entire study period, a median of 19.5 months
Population: No participants were enrolled in Groups CLL, CLL/BTK, CAR-T Cell and Other Adult Solid Tumor Booster Phase. Regarding Other Hematologic Malignancy Booster Phase Group 1 participant crossed over from hematologic low immunosuppression-initial phase; 3 participants crossed over from hematologic intermediate immunosuppression-initial phase; 3 participants crossed over from hematologic high immunosuppression-initial phase; & 3 participants were initially enrolled (did not cross over) into this group.
Measure: Count of Participants; unit: Participants
Groups:
- Chronic Lymphocytic Leukemia (CLL) Not on Active Therapy - Booster Phase; Chronic Lymphocytic Leukemia(CLL) Receiving Bruton´s Tyrosine Kinase(BTK) Interruption-Booster Phase; Chimeric Antigen Receptor (CAR) T Cell Therapy - Booster Phase; Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Booster Phase; Post Allogeneic Transplant - Booster Phase; Other Adult Solid Tumor - Booster Phase: 100 mcg (0.5 mL) messenger ribonucleic acid (mRNA)-1273 injection on day (D)1.
Arm/Group | Chronic Lymphocytic Leukemia (CLL) Not on Active Therapy - Booster Phase | Chronic Lymphocytic Leukemia(CLL) Receiving Bruton´s Tyrosine Kinase(BTK) Interruption-Booster Phase | Chimeric Antigen Receptor (CAR) T Cell Therapy - Booster Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Booster Phase | Post Allogeneic Transplant - Booster Phase | Other Hematologic Malignancy - Booster Phase | Other Adult Solid Tumor - Booster Phase
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 10 | 0
Participants
  Grade 1 Non-serious Solicited - Hemorrhoidal hemorrhage |  |  |  | 0 | 0 | 1 |
  Grade 1 Non-serious Solicited - Hypertension |  |  |  | 1 | 0 | 3 |
  Grade 1 Non-serious Solicited - Nasal congestion |  |  |  | 0 | 0 | 1 |
  Grade 1 Non-serious Solicited - Arthralgia |  |  |  | 0 | 0 | 1 |
  Grade 1 Non-serious Solicited - Weight gain |  |  |  | 0 | 1 | 0 |
  Grade 2 Non-serious Solicited - Conjunctivitis |  |  |  | 0 | 0 | 1 |
  Grade 2 Non-serious Solicited - Infections and infestations - Other COVID, specify |  |  |  | 0 | 1 | 3 |
  Grade 2 Non-serious Solicited - Neutrophil count decreased |  |  |  | 0 | 0 | 1 |
  Grade 2 Non-serious Solicited - Pneumonitis |  |  |  | 0 | 0 | 1 |
  Grade 2 Non-serious Solicited - Dental caries |  |  |  | 1 | 0 | 0 |
  Grade 2 Non-serious Solicited - Hypothyroidism |  |  |  | 1 | 0 | 0 |

4. Primary Outcome: Number of Participants Who Had Vital Signs Performed Prior to Vaccine
Description: Vital signs: weight, temperature, heart rate/pulse, respirations, and blood pressure will be performed prior to each vaccine.
Time Frame: Prior to each vaccine. Screening or Day 0 visit; Day 1, visit 1, vaccine dose 1; Day 29, visit 2, vaccine dose 2; Day 209 (6 months), visit 5 (+/- 28 days); and Day 394, visit 6 (+/- 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Hematologic Low Immunosuppression - Initial Phase | Hematologic Intermediate Immunosuppression - Initial Phase | Hematologic High Immunosuppression - Initial Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Initial Phase | Other Hematologic Malignancy - Booster Phase
Number analyzed (Participants) | 2 | 3 | 7 | 3 | 4
Participants
  Screening or Day 0 visit - Weight | 2 | 3 | 7 | 3 | 4
  Screening or Day 0 visit -Temperature | 2 | 3 | 7 | 3 | 4
  Screening or Day 0 visit - Heart rate/Pulse | 2 | 3 | 7 | 3 | 4
  Screening or Day 0 visit - Respirations | 2 | 3 | 7 | 3 | 4
  Screening or Day 0 visit - Blood Pressure | 2 | 3 | 7 | 3 | 4
  Day 1, visit 1, vaccine dose 1 - Weight | 2 | 3 | 7 | 3 | 0
  Day 1, visit 1, vaccine dose 1 - Temperature | 2 | 3 | 7 | 3 | 0
  Day 1, visit 1, vaccine dose 1 - Heart rate/Pulse | 2 | 3 | 7 | 3 | 0
  Day 1, visit 1, vaccine dose 1 - Respirations | 2 | 3 | 7 | 3 | 0
  Day 1, visit 1, vaccine dose 1 - Blood Pressure | 2 | 3 | 7 | 3 | 0
  Day 29, visit 2, vaccine dose 2 - Weight | 0 | 0 | 0 | 0 | 0
  Day 29, visit 2, vaccine dose 2 - Temperature | 2 | 3 | 6 | 3 | 0
  Day 29, visit 2, vaccine dose 2 - Heart rate/Pulse | 2 | 3 | 6 | 3 | 0
  Day 29, visit 2, vaccine dose 2 - Respirations | 2 | 3 | 6 | 3 | 0
  Day 29, visit 2, vaccine dose 2 - Blood Pressure | 2 | 3 | 6 | 3 | 0
  Day 209 (6 months), visit 5 (+/- 28 days) - Weight | 0 | 0 | 0 | 0 | 0
  Day 209 (6 months), visit 5 (+/- 28 days) - Temperature | 1 | 0 | 2 | 1 | 0
  Day 209 (6 months), visit 5 (+/- 28 days) - Heart rate/Pulse | 1 | 0 | 2 | 1 | 0
  Day 209 (6 months), visit 5 (+/- 28 days) - Respirations | 1 | 0 | 2 | 1 | 0
  Day 209 (6 months), visit 5 (+/- 28 days) - Blood Pressure | 1 | 0 | 2 | 1 | 0
  Day 394, visit 6 (+/- 28 days) - Weight | 0 | 0 | 0 | 0 | 0
  Day 394, visit 6 (+/- 28 days) - Temperature | 0 | 0 | 3 | 0 | 0
  Day 394, visit 6 (+/- 28 days) - Heart rate/Pulse | 0 | 0 | 3 | 0 | 0
  Day 394, visit 6 (+/- 28 days) - Respirations | 0 | 0 | 3 | 0 | 0
  Day 394, visit 6 (+/- 28 days) - Blood Pressure | 0 | 0 | 3 | 0 | 0

5. Primary Outcome: Immunogenicity of Messenger Ribonucleic Acid (mRNA) Titers - 1273 Administered in 2 Doses in the Initial Phase
Description: Immunogenicity of mRNA 1273 administered in 2 doses was assessed by titer or level of specific binding antibody (bAb), in participants who have a hematological malignancy and are immunosuppressed due to their disease and/or treatment or receiving a programmed death-1 (PD-1)/programmed death-ligand 1 inhibitor for treatment of a solid tumor - Titer or level of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)-specific binding antibody (bAb) measured by enzyme-linked immunosorbent assay (ELISA) on Day 1, Day 29, Day 36, Day 57, Day 209, and Day 394.
Time Frame: Day 1, Day 29, Day 36, Day 57, Day 209, and Day 394
Population: Day 394 Groups 1, 2 and 4 respectively; no participants reached this timepoint to be analyzed because, 1) the follow up was too short for participants and/or participants crossed over to the booster cohort.
Measure: Median (Full Range); unit: Au/mL
Units Other Than Participants: Blood samples
Arm/Group | Hematologic Low Immunosuppression - Initial Phase | Hematologic Intermediate Immunosuppression - Initial Phase | Hematologic High Immunosuppression - Initial Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Initial Phase
Number analyzed (Participants) | 2 | 3 | 7 | 3
Number analyzed (Blood samples) | 9 | 14 | 42 | 15
Au/mL
  Day 1: number analyzed (Blood samples) | 2 | 3 | 7 | 3
  Day 1 | 0 [0 to 0] | 0 [0 to 1.4] | 2.1 [0 to 815.2] | 0 [0 to 0.7]
  Day 29: number analyzed (Blood samples) | 2 | 3 | 7 | 3
  Day 29 | 0.3 [0 to 0.6] | 0 [0 to 8.4] | 838.4 [0.8 to 9276.0] | 608.3 [297.8 to 1982.4]
  Day 36: number analyzed (Blood samples) | 2 | 3 | 7 | 3
  Day 36 | 0.6 [0.1 to 1.2] | 0 [0 to 6.3] | 10830.2 [1.8 to 29849.1] | 35863.4 [26558.4 to 40941.6]
  Day 57: number analyzed (Blood samples) | 2 | 3 | 7 | 3
  Day 57 | 40.0 [39.2 to 40.7] | 0.23 [0 to 8.0] | 23084.7 [0.6 to 32795.2] | 27319.8 [20401 to 38429.7]
  Day 209: number analyzed (Participants) | 1 | 3 | 7 | 3
  Day 209: number analyzed (Blood samples) | 1 | 2 | 2 | 3
  Day 209 | 53156.4 [NA to 53156.4] — One out of two participants provided a sample, which was included for analysis. The other participant was not analyzed and moved to the booster cohort, so this timepoint was censored. | 53.7 [0 to 107.4] | 26153.9 [23639.6 to 28668.2] | 3198.9 [2467.1 to 4041.3]
  Day 394: number analyzed (Participants) | 0 | 0 | 7 | 0
  Day 394: number analyzed (Blood samples) | 0 | 0 | 3 | 0
  Day 394 |  |  | 24665.2 [20779.1 to 33967.9] |

6. Primary Outcome: Number of Participants With Reactogenicity of Messenger Ribonucleic Acid (mRNA) -1273 of a Booster Vaccination: Booster Phase
Description: Reactogenicity of mRNA-1273 of a booster vaccination was assessed by physical examination findings following vaccination. A physical exam will be performed to assess general physical condition in the following areas: supraclavicular and axillary lymph nodes, cardiovascular, pulmonary, abdomen and skin and include an assessment of pain, tenderness, erythema, induration and warmth at the injection site, fever, chills, arthralgia/joint pain, malaise/fatigue, myalgia/body aches, headache, nausea, vomiting, and abdominal pain following vaccination.
Time Frame: End of 15-minute observation period following each vaccination on Day 1 and Day 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Lymphocytic Leukemia (CLL) Not on Active Therapy - Booster Phase | Chronic Lymphocytic Leukemia(CLL) Receiving Bruton´s Tyrosine Kinase(BTK) Interruption-Booster Phase | Chimeric Antigen Receptor (CAR) T Cell Therapy - Booster Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Booster Phase | Post Allogeneic Transplant - Booster Phase | Other Hematologic Malignancy - Booster Phase | Other Adult Solid Tumor - Booster Phase
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 10 | 0
Participants
  Day 1 - Pain |  |  |  | 2 | 1 | 7 |
  Day 1 - Tenderness |  |  |  | 1 | 1 | 3 |
  Day 1 - Erythema |  |  |  | 2 | 0 | 2 |
  Day 1 - Induration and warmth at the injection site |  |  |  | 2 | 0 | 2 |
  Day 1 - Fever |  |  |  | 0 | 0 | 1 |
  Day 1 - Chills |  |  |  | 2 | 0 | 4 |
  Day 1 - Arthralgia/joint pain |  |  |  | 1 | 0 | 2 |
  Day 1 - Malaise/fatigue |  |  |  | 1 | 0 | 8 |
  Day 1 - Myalgia/body aches |  |  |  | 2 | 1 | 5 |
  Day 1 - Headache |  |  |  | 2 | 0 | 5 |
  Day 1 - Nausea |  |  |  | 0 | 0 | 2 |
  Day 1 - Vomiting |  |  |  | 0 | 0 | 0 |
  Day 1 - Abdominal pain |  |  |  | 0 | 0 | 0 |
  Day 29 - Pain |  |  |  | 0 | 0 | 2 |
  Day 29 - Tenderness |  |  |  | 0 | 0 | 1 |
  Day 29 - Erythema |  |  |  | 0 | 0 | 0 |
  Day 29 - Induration and warmth at the injection site |  |  |  | 0 | 0 | 0 |
  Day 29 - Fever |  |  |  | 0 | 0 | 0 |
  Day 29 - Chills |  |  |  | 0 | 0 | 0 |
  Day 29 - Arthralgia/joint pain |  |  |  | 0 | 0 | 0 |
  Day 29 - Malaise/fatigue |  |  |  | 0 | 0 | 0 |
  Day 29 - Myalgia/body aches |  |  |  | 0 | 0 | 1 |
  Day 29 - Headache |  |  |  | 0 | 0 | 1 |
  Day 29 - Nausea |  |  |  | 0 | 0 | 0 |
  Day 29 - Vomiting |  |  |  | 0 | 0 | 0 |
  Day 29 - Abdominal pain |  |  |  | 0 | 0 | 0 |

7. Secondary Outcome: Number of Neutralizing Antibody Samples - Initial Phase
Description: Number of samples with a neutralizing response (defined as neutralization assay above 30%) will be reported. Immunogenicity of mRNA-1273 vaccine was assessed for Vaccine Naive Arm in participants who have a hematological malignancy and are immunosuppressed due to their disease and/or treatment or receiving a programmed death-1 (PD-1)/programmed death-ligand 1 inhibitor for treatment of a solid tumor. Assessment was performed on Day 1, Day 29, Day 36, Day 57, Day 209, and Day 394
Time Frame: For Vaccine Naive Arm: Day 1, Day 29, Day 36, Day 57, Day 209, and Day 394
Population: as for outcome 5
Measure: Number; unit: Samples
Units Other Than Participants: Blood samples
Arm/Group | Hematologic Low Immunosuppression - Initial Phase | Hematologic Intermediate Immunosuppression - Initial Phase | Hematologic High Immunosuppression - Initial Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Initial Phase
Number analyzed (Participants) | 2 | 3 | 7 | 3
Number analyzed (Blood samples) | 9 | 14 | 33 | 15
Samples
  Day 1: number analyzed (Blood samples) | 2 | 3 | 7 | 3
  Day 1 | 0 | 0 | 2 | 0
  Day 29: number analyzed (Blood samples) | 2 | 3 | 7 | 3
  Day 29 | 0 | 0 | 5 | 3
  Day 36: number analyzed (Blood samples) | 2 | 3 | 7 | 3
  Day 36 | 0 | 0 | 6 | 3
  Day 57: number analyzed (Blood samples) | 2 | 3 | 7 | 3
  Day 57 | 0 | 0 | 6 | 3
  Day 209: number analyzed (Participants) | 1 | 2 | 2 | 3
  Day 209: number analyzed (Blood samples) | 1 | 2 | 2 | 3
  Day 209 | 1 | 1 | 2 | 3
  Day 394: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 394: number analyzed (Blood samples) | 0 | 0 | 3 | 0
  Day 394 |  |  | 3 |

8. Secondary Outcome: Number of Neutralizing Antibody Samples - Booster Phase
Description: Number of samples with a neutralizing response (defined as neutralization assay above 30%) will be reported. Participants would receive one to two vaccine boosters. Analysis of timepoints after booster 1 and booster 2 are reported collectively. Immunogenicity of mRNA-1273 vaccine was assessed for Booster Arm in participants with hematologic malignancy with or without ongoing immune suppression and participants with solid tumor receiving programmed death-1 (PD-1)/programmed death-ligand 1 inhibitor (PD-L1) inhibitors: Day 1, Day 29, Day 57, Day 180, and Day 360.
Time Frame: Day 1, Day 29, Day 57, Day 180, and Day 360
Population: as for outcome 3
Measure: Number; unit: Samples
Units Other Than Participants: Blood samples
Arm/Group | Chronic Lymphocytic Leukemia (CLL) Not on Active Therapy - Booster Phase | Chronic Lymphocytic Leukemia(CLL) Receiving Bruton´s Tyrosine Kinase(BTK) Interruption-Booster Phase | Chimeric Antigen Receptor (CAR) T Cell Therapy - Booster Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Booster Phase | Post Allogeneic Transplant - Booster Phase | Other Hematologic Malignancy - Booster Phase | Other Adult Solid Tumor - Booster Phase
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 10 | 0
Number analyzed (Blood samples) | 0 | 0 | 0 | 12 | 7 | 63 | 0
Samples
  Day 1: number analyzed (Blood samples) | 0 | 0 | 0 | 3 | 2 | 16 | 0
  Day 1 |  |  |  | 3 | 1 | 10 |
  Day 29: number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 9 | 0
  Day 29: number analyzed (Blood samples) | 0 | 0 | 0 | 3 | 2 | 15 | 0
  Day 29 |  |  |  | 3 | 2 | 12 |
  Day 57: number analyzed (Blood samples) | 0 | 0 | 0 | 3 | 1 | 13 | 0
  Day 57 |  |  |  | 3 | 1 | 10 |
  Day 180: number analyzed (Blood samples) | 0 | 0 | 0 | 2 | 1 | 10 | 0
  Day 180 |  |  |  | 2 | 1 | 10 |
  Day 360: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 9 | 0
  Day 360: number analyzed (Blood samples) | 0 | 0 | 0 | 1 | 1 | 9 | 0
  Day 360 |  |  |  | 1 | 1 | 9 |

9. Secondary Outcome: Immunogenicity of Messenger Ribonucleic Acid (mRNA) -1273 Levels Administered in 2 Doses in the Booster Phase
Description: Immunogenicity of mRNA 1273 administered in 2 doses was assessed by titer or level of specific binding antibody (bAb), in participants with hematologic malignancy with or without ongoing immune suppression and patients with solid tumor receiving programmed death-1 (PD-1)/programmed death-ligand 1 inhibitor (PD-L1) inhibitors. Titer or level of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)-specific binding antibody (bAb) measured by enzyme-linked immunosorbent assay (ELISA) on Day 1, Day 29, Day 57, Day 180, and Day 360. Participants received one or two vaccine boosters. Analysis of timepoints after booster 1 and booster 2 are reported collectively.
Time Frame: Day 1, Day 29, Day 57, Day 180, and Day 360
Population: as for outcome 3
Measure: Median (Full Range); unit: AU/mL
Units Other Than Participants: Blood samples
Arm/Group | Chronic Lymphocytic Leukemia (CLL) Not on Active Therapy - Booster Phase | Chronic Lymphocytic Leukemia(CLL) Receiving Bruton´s Tyrosine Kinase(BTK) Interruption-Booster Phase | Chimeric Antigen Receptor (CAR) T Cell Therapy - Booster Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Booster Phase | Post Allogeneic Transplant - Booster Phase | Other Hematologic Malignancy - Booster Phase | Other Adult Solid Tumor - Booster Phase
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 10 | 0
Number analyzed (Blood samples) | 0 | 0 | 0 | 12 | 7 | 63 | 0
AU/mL
  Day 1: number analyzed (Blood samples) | 0 | 0 | 0 | 3 | 2 | 16 | 0
  Day 1 |  |  |  | 4041.3 [3198.9 to 18374.8] | 23271.4 [0 to 46542.7] | 4904.71 [0 to 39676.1] |
  Day 29: number analyzed (Blood samples) | 0 | 0 | 0 | 3 | 2 | 15 | 0
  Day 29 |  |  |  | 30161.9 [19237.6 to 44659.6] | 43021.6 [39500.5 to 46542.7] | 22317.0 [0 to 52133.4] |
  Day 57: number analyzed (Blood samples) | 0 | 0 | 0 | 3 | 1 | 13 | 0
  Day 57 |  |  |  | 45003.9 [33714.8 to 49317.2] | 32364.0 [upper limit 32364.0] | 16527.2 [0 to 33450.0] |
  Day 180: number analyzed (Blood samples) | 0 | 0 | 0 | 2 | 1 | 10 | 0
  Day 180 |  |  |  | 18918.0 [10902.5 to 26933.5] | 10662.5 [upper limit 10662.5] | 11842.9 [1594.0 to 38181.6] |
  Day 360: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 10 | 0
  Day 360: number analyzed (Blood samples) | 0 | 0 | 0 | 1 | 1 | 9 | 0
  Day 360 |  |  |  | 22329.9 [NA to 22329.9] — One out of two participants and one sample analyzed here. | 2331.7 [NA to 2331.7] — One sample analyzed here. | 8555.06 [1855.4 to 114586.3] |

10. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: From study product administration on Day 1 through 28 days after the last vaccination (through resolution); a median of 19.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Hematologic Low Immunosuppression - Initial Phase | Hematologic Intermediate Immunosuppression - Initial Phase | Hematologic High Immunosuppression - Initial Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Initial Phase | Other Hematologic Malignancy - Booster Phase
Number analyzed (Participants) | 2 | 3 | 7 | 3 | 4
Participants | 2 | 1 | 6 | 2 | 3

ADVERSE EVENTS:
Time Frame: From study product administration on Day 1 through 28 days after the last vaccination (through resolution); a median of 19.5 months.
Arm/Group | Hematologic Low Immunosuppression - Initial Phase | Hematologic Intermediate Immunosuppression - Initial Phase | Hematologic High Immunosuppression - Initial Phase | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Initial Phase | Other Hematologic Malignancy - Booster Phase
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/7 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 2/7 | 1/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2/2 | 1/3 | 6/7 | 2/3 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematologic Low Immunosuppression - Initial Phase (N=2) | Hematologic Intermediate Immunosuppression - Initial Phase (N=3) | Hematologic High Immunosuppression - Initial Phase (N=7) | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Initial Phase (N=3) | Other Hematologic Malignancy - Booster Phase (N=4)
Immune system disorders - Other, Graft versus host disease (GVHD) (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematologic Low Immunosuppression - Initial Phase (N=2) | Hematologic Intermediate Immunosuppression - Initial Phase (N=3) | Hematologic High Immunosuppression - Initial Phase (N=7) | Solid Tumor on Programmed Cell Death protein1/Programmed Cell Death Ligand 1 Inhibitor-Initial Phase (N=3) | Other Hematologic Malignancy - Booster Phase (N=4)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune system disorders - Other, chronic graft vs. host disease (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) — Includes body aches, headache, fever, dry cough
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, COVID-19 infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Gastrointestinal (GI) virus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT04847050/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT04847050/ICF_001.pdf